CLINICAL TRIAL: NCT05783791
Title: Development of a Newborn Screening Assay for Angelman Syndrome and Prader-Willi Syndrome
Status: Completed | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Ultragenyx Pharmaceutical Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: 2022-1467; WSLH Newborn Screening (Other: UW Madison); CP001 approved 1/31/2023 (Other: UW Madison)
Record Dates: First submitted 2023-03-13; First posted 2023-03-24 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-08

CONDITIONS: Angelman Syndrome; Prader-Willi Syndrome
Keywords: Newborn Screening; Assay; Public Health
MeSH Terms: conditions — Angelman Syndrome; Prader-Willi Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

GROUPS / COHORTS (3):
- Participants with Angelman Syndrome (AS): AS confirmed by molecular testing
  Interventions: Diagnostic Test: Newborn Screening Assay
- Participants with Prader-Willi Syndrome (PWS): PWS confirmed by molecular testing
  Interventions: Diagnostic Test: Newborn Screening Assay
- Healthy Controls
  Interventions: Diagnostic Test: Newborn Screening Assay

INTERVENTIONS:
Diagnostic Test: Newborn Screening Assay — The assay developed in this study is determined to be FDA regulated as an exempt diagnostic device. In this study, the testing involved with this assay fulfills the following criteria:
  * Is noninvasive
  * Does not require an invasive sampling procedure that presents significant risk (the finger prick is minimal risk)
  * Does not by design or intention introduce energy into a subject, and
  * Is not used as a diagnostic procedure without confirmation of the diagnosis by another, medically established diagnostic product or procedure, as participants will not receive results in this study.

SUMMARY:
The overall purpose of this project is to establish the capability of screening for Angelman syndrome (AS) and Prader-Willi syndrome (PWS) in public health newborn screening (NBS) programs, with an aim of developing and validating a screening test for AS and PWS.

DETAILED DESCRIPTION:
This project will have an assay development phase and an assay validation phase.

In the assay development phase, the investigators will develop a method of assessing SNRPN promoter (located in chromosome 15 q11-q13) methylation status using methylation-specific PCR coupled with a melting curve analysis with de-identified leftover DNA from routine newborn screening dried blood samples for severe combined immunodeficiency and spinal muscular atrophy.

In the assay validation phase, the investigators plan to assess the assay sensitivity and specificity using a set of DNA samples extracted from dried blood spots in each following group:

1. Healthy individuals
2. AS patients with genetic testing confirmation that the maternal copy of chromosome 15 q11-q13 is deleted, or that there are two paternal copies of chromosome 15 q11-q13 or imprinting center defect.
3. PWS patients with genetic testing confirmation that the paternal copy of chromosome 15 q11-q13 is deleted, or that there are two maternal copies of chromosome 15 q11-q13 or imprinting center defect.

For participants with AS or PWS, blood samples will be obtained via a self-administered finger prick performed in the participant's home. The participant will mail the sample to the researchers using a provided envelope. If the team is not able to reach the participant after two phone call attempts, the study team may approach them at their next clinic visit to assess interest in study participation. If participants opt to join the study at this clinic visit, the blood sample may be obtained in clinic.

For healthy controls, blood samples will be obtained via a self-administered finger prick, and participants will verbally respond to a brief demographic questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Angelman Syndrome, confirmed by molecular testing (deletion of maternal allele of chromosome 15q11-q13, paternal uniparental disomy, and imprinting center defects)
* Diagnosed with Prader-Willi Syndrome, confirmed by molecular testing (deletion of paternal allele of chromosome 15q11-q13, maternal uniparental disomy, and imprinting center defects)
* Angelman Syndrome or Prader Willi Syndrome: Current patient at UW Health in the Madison, Wisconsin metropolitan area
* Healthy controls 18 years old or older and have not received a diagnosis of Angelman syndrome or Prader Willi syndrome

Exclusion Criteria:

* Angelman Syndrome/Prader Willi Syndrome: family requires a translator for medical visits
* Healthy Controls: Participants are unable to consent and complete study procedures in English.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: This study will target three groups:
  * participants with Angelman Syndrome
  * participants with Prader-Willi Syndrome
  * healthy controls
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2023-04-20 (Actual); Primary Completion 2023-07-21 (Actual); Study Completion 2023-07-21 (Actual)

PRIMARY OUTCOMES:
Sensitivity: Number of True Positive AS Results | 1 sample collected from participant either at home or in presence of a study team member at clinic, up to 5 minutes
Sensitivity: Number of True Positive PWS Results | 1 sample collected from participant either at home or in presence of a study team member at clinic, up to 5 minutes
Specificity: Number of Healthy Controls With True Negative Results | 1 sample collected from participant in presence of a study team member (controls), up to 5 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Mei W Baker, M.D., FACMG, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin School of Medicine and Public Health, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2023-01-23): https://cdn.clinicaltrials.gov/large-docs/91/NCT05783791/ICF_000.pdf